CLINICAL TRIAL: NCT02275637
Title: Arrhythmias Detection in a Real World Population: the RHYTHM DETECT Registry
Brief Title: Arrhythmias Detection in a Real World Population
Acronym: RHYTHM DETECT
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Maurizio Eugenio Landolina, EP and Pacing Laboratory Director, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 20140002277 del 27/05/2014
Record Dates: First submitted 2014-10-09; First posted 2014-10-27 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-01

CONDITIONS: Appropriate and Inappropriate Shock Therapy With ICD; Arrhythmias Detection
Keywords: Implantable Cardioverter-Defibrillators; Ventricular Fibrillation; ventricular Tachycardia
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: implantable cardioverter defibrillator

SUMMARY:
The study is a prospective multicenter registry. Consecutive patients with indications of implant / replacement or upgrade of implantable cardioverter defibrillator (ICD) will be enrolled.

The primary objective of the study is to determine the predictors of appropriate anti-tachycardia therapy (with shock) in a non-selected population of patients implanted with an ICD.

Secondary objectives of the study are:

* the incidence of anti-tachycardia therapies;
* the predictors of inappropriate therapy and onset of arrhythmia burden;
* the adherence to the current guidelines in the Italian clinical practice;
* the predictors of heart failure (HF) onset and response to cardiac resynchronization therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with a Subcutaneous (S)- Ventricular Chamber (VR)- Dual Chamber (DR) - or Cardiac Resynchronization Therapy (CRT) Defibrillator (this study will utilize all the market released CRT-D or VR/DR-ICD systems and leads)
* Patient is willing and able to sign an authorization to use and disclose health information or an Informed Consent
* Patient must be able to attend all required follow-up visits at the study center for at least 12 months

Exclusion Criteria:

* Patient is participating in another clinical study that may have an impact on the study endpoints
* Women who are pregnant or plan to become pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study requires patients implanted with a defibrillator that meet all inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-09; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patients with ICD therapy (shock) | 24 months
  Clinical or instrumental parameters that could predict the appropriate ICD therapies

SECONDARY OUTCOMES:
Patients with inappropriate shock therapy | 24 months
  Clinical or instrumental parameters that could predict the inappropriate ICD therapies
Incidence of ICD therapies | 24 months
  Number of patients with ICD therapies
Time to first ICD therapy | 24 months
Predictors of onset and Atrial Fibrillation (AF) burden | 24 months

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Policlinico S.Orsola-Malpighi, Bologna
  - P.O. Rodolico-San Marco, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - ASST Rhodense- Ospedale di Rho, Milan
  - IRCCS S.Ambrogio-Galeazzi, Milan
  - Ospedale dei Colli Monaldi, Naples
  - University of Padua, Padua
  - IRCC Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisa Cisanello, Pisa
  - Azienda Ospedaliera S.Andrea, Rome
  - Ospedale Bambino Gesù, Rome

REFERENCES:
- [Derived] Migliore F, Ottaviano L, Arestia A, Nigro G, Dello Russo A, Viani S, Bianchi V, Bisignani A, Pieragnoli P, Vitulano G, Rordorf R, Francia P, Taravelli E, Pisano E, Lavalle C, Brambilla R, Ziacchi M, Rapacciuolo A, Viscusi M, De Filippo P, La Greca C, Pepi P, Notarstefano P, Curcio A, Pittorru R, Martini N, Seganti A, Napolitano C, Lovecchio M, Valsecchi S, Botto G, Priori SG; S-ICD Rhythm Detect Investigators. Subcutaneous Implantable Defibrillator Therapy in Patients With Brugada Syndrome: Data From a Large Multicenter Registry. JACC Clin Electrophysiol. 2025 Jul;11(7):1572-1582. doi: 10.1016/j.jacep.2025.03.003. Epub 2025 Mar 29. PMID 40156599
- [Derived] Ziacchi M, Ottaviano L, Checchi L, Viani S, Nigro G, Bianchi V, De Bonis S, De Filippo P, Francia P, Rapacciuolo A, Vitulano G, Perego GB, Schillaci V, Lavalle C, Migliore F, Pisano ECL, Compagnucci P, Palmisano P, Botto G, Rordorf R, Lovecchio M, Valsecchi S, Biffi M. The risk of failure of subcutaneous implantable cardioverter defibrillator therapy: from PRAETORIAN score to clinical practice. Europace. 2025 Feb 5;27(2):euaf011. doi: 10.1093/europace/euaf011. PMID 39834232
- [Derived] Boriani G, Bertini M, Manzo M, Calo L, Santini L, Savarese G, Dello Russo A, Santobuono VE, Lavalle C, Viscusi M, Amellone C, Calvanese R, Santoro A, Rapacciuolo A, Ziacchi M, Arena G, Imberti JF, Campari M, Valsecchi S, D'Onofrio A. Performance of a multi-sensor implantable defibrillator algorithm for heart failure monitoring in the presence of atrial fibrillation. Europace. 2023 Aug 2;25(9):euad261. doi: 10.1093/europace/euad261. PMID 37656991
- [Derived] Migliore F, Biffi M, Viani S, Pittorru R, Francia P, Pieragnoli P, De Filippo P, Bisignani G, Nigro G, Dello Russo A, Pisano E, Palmisano P, Rapacciuolo A, Silvetti MS, Lavalle C, Curcio A, Rordorf R, Lovecchio M, Valsecchi S, D'Onofrio A, Botto GL. Modern subcutaneous implantable defibrillator therapy in patients with cardiomyopathies and channelopathies: data from a large multicentre registry. Europace. 2023 Aug 2;25(9):euad239. doi: 10.1093/europace/euad239. PMID 37536671
- [Derived] De Filippo P, Migliore F, Palmisano P, Nigro G, Ziacchi M, Rordorf R, Pieragnoli P, Di Grazia A, Ottaviano L, Francia P, Pisano E, Tola G, Giammaria M, D'Onofrio A, Botto GL, Zucchelli G, Ferrari P, Lovecchio M, Valsecchi S, Viani S. Procedure, management, and outcome of subcutaneous implantable cardioverter-defibrillator extraction in clinical practice. Europace. 2023 Jun 2;25(6):euad158. doi: 10.1093/europace/euad158. PMID 37350404
- [Derived] Santobuono VE, Favale S, D'Onofrio A, Manzo M, Calo L, Bertini M, Savarese G, Santini L, Dello Russo A, Lavalle C, Viscusi M, Amellone C, Calvanese R, Arena G, Pangallo A, Rapacciuolo A, Porcelli D, Campari M, Valsecchi S, Guaricci AI. Performance of a multisensor implantable defibrillator algorithm for heart failure monitoring related to co-morbidities. ESC Heart Fail. 2023 Aug;10(4):2469-2478. doi: 10.1002/ehf2.14416. Epub 2023 Jun 5. PMID 37278122
- [Derived] Rordorf R, Viani S, Biffi M, Pieragnoli P, Migliore F, D'Onofrio A, Nigro G, Francia P, Ferrari P, Dello Russo A, Bisignani A, Ottaviano L, Palmisano P, Caravati F, Pisano E, Pani A, Botto GL, Lovecchio M, Valsecchi S, Vicentini A. Reduction in inappropriate therapies through device programming in subcutaneous implantable defibrillator patients: data from clinical practice. Europace. 2023 May 19;25(5):euac234. doi: 10.1093/europace/euac234. PMID 36932709
- [Derived] Bertini M, Vitali F, D'Onofrio A, Vitulano G, Calo L, Savarese G, Santobuono VE, Dello Russo A, Mattera A, Santoro A, Calvanese R, Arena G, Amellone C, Ziacchi M, Palmisano P, Santini L, Mazza A, Campari M, Valsecchi S, Boriani G. Combination of an implantable defibrillator multi-sensor heart failure index and an apnea index for the prediction of atrial high-rate events. Europace. 2023 Apr 15;25(4):1467-1474. doi: 10.1093/europace/euad052. PMID 36881780
- [Derived] Botto GL, Ziacchi M, Nigro G, D'Onofrio A, Dello Russo A, Francia P, Viani S, Pisano E, Bisignani G, Caravati F, Migliore F, De Filippo P, Ottaviano L, Rordorf R, Manzo M, Canevese FL, Lovecchio M, Valsecchi S, Checchi L. Intermuscular technique for implantation of the subcutaneous implantable defibrillator: a propensity-matched case-control study. Europace. 2023 Apr 15;25(4):1423-1431. doi: 10.1093/europace/euad028. PMID 36794691
- [Derived] Mazza A, Bendini MG, Bianchi V, Esposito C, Calo L, Andreoli C, Santobuono VE, Dello Russo A, Viscusi M, La Greca C, Baiocchi C, Talarico A, Albanese R, Arena G, Giubilato G, Ziacchi M, Rapacciuolo A, Campari M, Valsecchi S, Boriani G. Association Between Device-Detected Sleep-Disordered Breathing and Implantable Defibrillator Therapy in Patients With Heart Failure. JACC Clin Electrophysiol. 2022 Oct;8(10):1249-1256. doi: 10.1016/j.jacep.2022.07.017. Epub 2022 Sep 28. PMID 36266001
- [Derived] Vicentini A, Bisignani G, De Vivo S, Viani S, Savarese G, Francia P, Celentano E, Checchi L, Carreras G, Santini L, Lamberti F, Ottaviano L, Scalone A, Giorgi D, Lovecchio M, Valsecchi S, Rordorf R; "S-ICD Rhythm Detect" Investigators. Patient acceptance of subcutaneous versus transvenous defibrillator systems: A multi-center experience. J Cardiovasc Electrophysiol. 2022 Jan;33(1):81-89. doi: 10.1111/jce.15297. Epub 2021 Nov 28. PMID 34797012
- [Derived] Russo V, Viani S, Migliore F, Nigro G, Biffi M, Tola G, Bisignani G, Dello Russo A, Sartori P, Rordorf R, Ottaviano L, Perego GB, Checchi L, Segreti L, Bertaglia E, Lovecchio M, Valsecchi S, Bongiorni MG. Lead Abandonment and Subcutaneous Implantable Cardioverter-Defibrillator (S-ICD) Implantation in a Cohort of Patients With ICD Lead Malfunction. Front Cardiovasc Med. 2021 Jul 27;8:692943. doi: 10.3389/fcvm.2021.692943. eCollection 2021. PMID 34395560
- [Derived] Calo L, Bianchi V, Ferraioli D, Santini L, Dello Russo A, Carriere C, Santobuono VE, Andreoli C, La Greca C, Arena G, Talarico A, Pisano E, Santoro A, Giammaria M, Ziacchi M, Viscusi M, De Ruvo E, Campari M, Valsecchi S, D'Onofrio A; Full list of participant centers and investigators. Multiparametric Implantable Cardioverter-Defibrillator Algorithm for Heart Failure Risk Stratification and Management: An Analysis in Clinical Practice. Circ Heart Fail. 2021 Oct;14(10):e008134. doi: 10.1161/CIRCHEARTFAILURE.120.008134. Epub 2021 Jun 30. PMID 34190592
- [Derived] Francia P, Adduci C, Angeletti A, Ottaviano L, Perrotta L, De Vivo S, Bongiorni MG, Migliore F, Russo AD, De Filippo P, Caravati F, Nigro G, Palmisano P, Viani S, D'Onofrio A, Lovecchio M, Valsecchi S, Ziacchi M. Acute shock efficacy of the subcutaneous implantable cardioverter-defibrillator according to the implantation technique. J Cardiovasc Electrophysiol. 2021 Jun;32(6):1695-1703. doi: 10.1111/jce.15081. Epub 2021 May 16. PMID 33969578
- [Derived] Francia P, Biffi M, Adduci C, Ottaviano L, Migliore F, De Bonis S, Dello Russo A, De Filippo P, Viani S, Bongiorni MG, Caravati F, Lavalle C, Landolina ME, Pisano E, Giorgi D, Lovecchio M, Valsecchi S, Diemberger I. Implantation technique and optimal subcutaneous defibrillator chest position: a PRAETORIAN score-based study. Europace. 2020 Dec 23;22(12):1822-1829. doi: 10.1093/europace/euaa231. PMID 33118017
- [Derived] Ziacchi M, Bisignani G, Palmisano P, Scalone A, Martignani C, Elvira Mocavero P, Caravati F, Della Cioppa N, Mazzuero A, Pecora D, Vicentini A, Landolina ME, Debonis S, Scimia P, Lovecchio M, Valsecchi S, Diemberger I, Droghetti A. Serratus anterior plane block in subcutaneous implantable cardioverter defibrillator implantation: A case-control analysis. J Cardiovasc Electrophysiol. 2020 Jan;31(1):144-149. doi: 10.1111/jce.14293. Epub 2019 Dec 3. PMID 31778266
- [Derived] Diemberger I, Migliore F, Ricciardi G, Ottaviano L, Tavoletta V, Francia P, Viani S, Capucci A, de Filippo P, Nigro G, Caravati F, Palmisano P, Ziacchi M, Lovecchio M, Valsecchi S, Bongiorni MG, Biffi M; "S-ICD Rhythm Detect" Investigators. Time to therapy delivery and effectiveness of the subcutaneous implantable cardioverter-defibrillator. Heart Rhythm. 2019 Oct;16(10):1531-1537. doi: 10.1016/j.hrthm.2019.05.028. Epub 2019 May 29. PMID 31150817